CLINICAL TRIAL: NCT02200861
Title: Tooth Extraction With Deep Sedation in Children: A Retrospective Study
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Dilek Günay CANPOLAT, Associate Professor, TC Erciyes University
Other Study IDs: 2014/389
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Tooth Extraction Status Nos
Keywords: sedation,; tooth extraction,

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study it's aimed to evaluated the patients in whom dental local anesthetic attempts were failed due to anxiety or fear and referred to our clinic for tooth extraction with deep sedation. All patients dates will evaluate from their patient file retrospectively from 2011 to 2014.

DETAILED DESCRIPTION:
Majority of dental treatments can be performed under local anesthesia. However, this is not always possible for pediatric non-cooperated patients with severe anxiety. In these patients, unpleasant dental experiences may lead to development of dental phobia when they become adults . Therefore, it is important to eradicate anxiety, and to prevent a possible psychological trauma in pediatric patients. For this purpose, psychological and medical methods have been applied to increase patient compliance. It has been proven that general anesthesia especially prevents dental phobia in elderly, and increases the quality of life related to oral health. In this study we aimed to evaluated the patients in whom dental local anesthetic attempts were failed due to anxiety or fear and referred to our clinic for tooth extraction with deep sedation. All patients dates will evaluate from their patient file retrospectively from 2011 to 2014.

ELIGIBILITY:
Inclusion Criteria:

* the patients who dental treatment was performed with deep sedation

Exclusion Criteria:

* the patients who dental treatment was performed local anesthesia or general anesthesia

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children
Sampling Method: Probability Sample
Enrollment: 885 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
anesthetic technics used for deep sedation | 2 month

SECONDARY OUTCOMES:
side effects observed in patients | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)